CLINICAL TRIAL: NCT05134246
Title: Outcomes of Carotid Revascularization for Patients With Radiation Induced Carotid Artery Stenosis in China
Brief Title: Carotid Revascularization for Radiation Induced Carotid Artery Stenosis
Acronym: CRICS
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CRICS
Record Dates: First submitted 2021-11-11; First posted 2021-11-24 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Radiation-induced Carotid Artery Stenosis
Keywords: Radiation-induced carotid artery stenosis; Carotid endarterectomy; Outcomes
MeSH Terms: interventions — Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — We will collect the carotid plaque for patients treated with carotid endarterectomy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Carotid endarterectomy (CEA): Patients who are treated with CEA.
  Interventions: Procedure: Carotid endarterectomy (CEA)
- Carotid artery stenting (CAS): Patients who are treated with CAS.
  Interventions: Procedure: Carotid artery stenting (CAS)

INTERVENTIONS:
Procedure: Carotid endarterectomy (CEA) — Surgeons follow the contemporary guideline combined with their experience and preference in order to ultimately select what is best suited for the patient and choose between CEA and CAS. Patients will receive 100 mg of aspirin or 75 mg of clopidogrel daily starting from at least 72 h prior to the CEA procedure and continued receiving the medication indefinitely. General anesthesia is recommended for CEA, although the use of standard or eversion endarterectomy, and a shunt or patch, is left to the discretion of the surgeon.
  Groups: Carotid endarterectomy (CEA)
Procedure: Carotid artery stenting (CAS) — Surgeons follow the contemporary guideline combined with their experience and preference in order to ultimately select what is best suited for the patient and choose between CEA and CAS. Patients will be given 100 mg of aspirin plus 75 mg of clopidogrel daily for at least 3 days before the CAS procedure and for 90 days after the procedure. They will receive a daily dose of 100 mg aspirin or 75 mg clopidogrel thereafter. For the CAS procedure, local anaesthesia and predilation prior to stent placement are recommended. Use of an embolic protection device is mandatory for all patients who undergo CAS.
  Groups: Carotid artery stenting (CAS)

SUMMARY:
Cervical radiotherapy (RT) has greatly reduced the mortality of patients with malignant head and neck tumors, which, however, causes a higher risk of carotid artery stenosis, namely, radiation-induced carotid artery stenosis (RICS) and results in a significant increased risk of ischemic stroke. The systematic review and meta-analysis conducted by our team showed carotid endarterectomy (CEA) can yield better results for these patients than carotid artery stenting (CAS), which was contrary to most previous clinical guidelines. A large-scale prospective study is needed to verify the results. We will conduct a prospective registry of RICS patients treated with CEA to evaluate both short-term safety and long-term efficacy outcomes in a Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with carotid stenosis who had a history of radiotherapy for head and neck cancer. (The median interval between the completion of radiation therapy and development of carotid artery stenosis detected on imaging (or vascular intervention) was no less than 1 years to avoid non-related situations. The target area of the radiotherapy included at least the ipsilateral neck, including part of the carotid system. The internal carotid stenosis was confirmed by angiography, Duplex, 3D angio-CTA or angio-MRI, and stenosis was defined as > 50% based on North American Symptomatic Carotid Endarterectomy Trial criteria), with or without symptom. Patients with a transient ischaemic attack (TIA) or stroke within 6 months were defined as symptomatic. TIA was defined as a transient episode of neurological dysfunction (focal weakness/ language disturbance/transient monocular blindness/ requiring assistance to walk) caused by focal brain or retinal ischemia that lasts for at least 10 min but resolves within 24 h.)

Exclusion Criteria:

* The patients treated for restenosis.
* Intracranial arteriovenous malformation or aneurysm
* Severe stenosis or occlusion of the ipsilateral intracranial artery
* Unstable angina, myocardial infarction (MI), or congestive heart failure in the last 6 months
* Uncorrectable coagulation abnormalities
* Uncontrolled diabetes mellitus defined as glucose > 300 mg/dL (16.67 mmol/L)
* Pregnant or in the perinatal period
* Severe concomitant disease with poor prognosis (life expectancy < 2 years)
* Intolerance or allergies to any of the study medications, such as aspirin or clopidogrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with RICS and fulfilled the above eligible criteria in tertiary medical centers in China, will be enrolled consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-01-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Stroke or death within 1 month | Within 1-month post-procedure
  A composite of any stroke or death occurring within 1-month post-procedure.

SECONDARY OUTCOMES:
Stroke beyond 1 month within 1 year | Beyond 1-month and within 1 year post-procedure
  Stroke beyond 1 month within 1 year
Death beyond 1 month within 1 year | Beyond 1-month and within 1 year post-procedure
  Death beyond 1 month within 1 year
Stroke or death within 1 year | Within 1 year post-procedure
  Stroke or death within 1 year
Cranial nerve injury | Within 1-month post-procedure
  Number of participants who suffered from cranial nerve injury
Carotid artery restenosis | Within 1-year post-procedure
  Number of participants who suffered from carotid artery restenosis (> 50%) detected by ultrasonography, CTA, or DSA
Functional outcome | Within 1-year post-procedure
  Functional outcome indicated by NIHSS (National Institutes of Health Stroke Scale: 0-42; higher scores indicate worse outcome) or mRS (modified Rankin Scale: 0-6; higher scores indicate worse outcome)
Other major complications | Within 1-month post-procedure
  Other major complications, such as myocardial infarction, incision hematoma, pulmonary infection, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Liqun Jiao, MD, Study Chair — Xuanwu Hospital, Beijing; Tao Wang, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (2):
- China (2):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided
Please contact the PI.